CLINICAL TRIAL: NCT04935216
Title: Predictors of Postoperative Complications and Readmissions in Laparoscopic Pancreas Resection: Results of 105 Consecutive Cases
Brief Title: Predictors of Postoperative Complications and Readmissions in Laparoscopic Pancreas Resection
Status: Completed | Type: Observational
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Other Study IDs: LAPAN
Record Dates: First submitted 2021-05-07; First posted 2021-06-22 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Laparoscopic Surgery; Pancreas
MeSH Terms: interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Laparoscopic — Laparoscopic resection of the pancreas has become widely accepted in the treatment of lesions which are benign or of low-grade malignancy

SUMMARY:
Laparoscopic resection of the pancreas has become widely accepted in the treatment of lesions which are benign or of low-grade malignancy. The objective of this study is to analyze the factors that predict postoperative complications and hospital readmission in a series of laparoscopic pancreatectomies.

DETAILED DESCRIPTION:
The investigators conducted a retrospective study using a prospective database of laparoscopic resections performed between 2000 and 2020. Data were collected on age, gender, body mass index (BMI), American Society of Anesthesiology (ASA) score, type of surgery, histologic type, operative time, hospital stay, postoperative complications, degree of severity and hospital readmission

ELIGIBILITY:
Inclusion Criteria:

* A retrospective study was carried out using data from a prospective database of all consecutive patients undergoing laparoscopic resection of the pancreas between 2000 and 2020 in the Clínica Universidad de Navarra

Exclusion Criteria:

* n/a

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients undergoing laparoscopic resection of the pancreas between 2000 and 2020 in the Clínica Universidad de Navarra
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2000-01 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Correlation of Gender, Age, body mass index with the outcomes | 20 years
  The investigators evaluate multiple variables in relation in the designed outcomes: Gender, Age, body mass index (weight and height will be combined to report BMI in kg/m^2)
Readmission | 60 days
  Readmission defined as an admission to any hospital for 24 hours or more for any reason within 60 days of surgery

IPD SHARING:
Plan to Share IPD: No